CLINICAL TRIAL: NCT00820365
Title: Exploratory, Open-label Study to Demonstrate Efficacy, Safety and Tolerability of SC12267 (35 mg) in Patients With Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis)
Brief Title: SC12267 (4SC-101) for Treatment of Patients With Inflammatory Bowel Disease
Acronym: ENTRANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 4SC AG (Industry)
Responsible Party: Dr. Bernhard Hauns, Medical Director Oncology, 4SC AG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC12267-4-2008; EudraCT-Number: 2008-005903-25
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Inflammatory Bowel Disease (IBD); Crohn's Disease; Ulcerative Colitis; SC12267; 4SC-101; Phase II
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — vidofludimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SC12267 (4SC-101) — Peroral administration of SC12267 (4SC-101) in patients with Inflammatory Bowel Disease over 12 weeks.

SUMMARY:
This is an exploratory, open-label, uncontrolled, multi-center, 1-arm study conducted at 16 sites in Bulgaria, Germany and Romania.

A total of ca. 30 - 35 patients will receive SC12267 (4SC-101) tablets, 35 mg once daily for 12 weeks. First of all the patients will undergo a screening period of 1 week and a follow-up visit will be performed 4 weeks after study drug discontinuation or earlier in case of relapse during follow up. Total study duration will be up to 36 (+2) weeks.

There will be 8 study visits: one screening visit, 6 visits during the treatment period and one follow-up visit. In addition, four telephone visits will be performed at Week 6, Week 10, Week 20 (+1) and Week 36 (+2).

The duration of the entire study (first patient in till last patient out) is expected to be about 13 months.

ELIGIBILITY:
Inclusion Criteria:

Criteria regarding Crohn´s Disease:

* Established diagnosis of CD, confirmed by standard criteria (e.g. endoscopy, ultrasound, X-ray)
* Patients must be in clinical remission (Crohn's Disease Activity Index [CDAI] <150 points) on steroid therapy for at least 2 weeks
* Confirmed steroid-dependency of CD: patients who are either

  1. unable to taper steroids completely within 3 months of starting steroids, without recurrent active disease, or
  2. who have a relapse within 2 months of stopping steroids
* Individual threshold* dose of previous relapses should be equal or less than 20 mg/day Prednisolone or equivalent steroid dose
* Patients with stable glucocorticosteroid therapy between 20 and 40 mg/day Prednisolone or equivalent steroid dose for the previous week

Criteria regarding Ulcerative Colitis:

* Established diagnosis of UC, confirmed by standard criteria (e.g. endoscopy, ultrasound, X-ray)
* Patients must be in clinical remission (Clinical Activity Index [CAI] <4 points) on steroid therapy for at least 2 weeks
* Confirmed steroid-dependency of UC: patients who are either

  1. unable to taper steroids completely within 3 months of starting steroids, without recurrent active disease, or
  2. who have a relapse within 2 months of stopping steroids
* Individual threshold* dose of previous relapses should be equal or less than 20 mg/day Prednisolone or equivalent steroid dose
* Patients with stable glucocorticosteroid therapy between 20 and 40 mg/day Prednisolone or equivalent steroid dose for the previous week

(* The threshold dose is that dose at which the patient experienced the relapses)

Criteria regarding general requirements:

* Men and women, 18 to 70 years of age
* Written informed consent
* Negative pregnancy test at screening in females of child-bearing potential
* Males willing to use condoms or to be sexually abstinent
* Use of appropriate contraceptive methods for females of childbearing potential one month before, throughout the course of the study and one month after study termination. This must be a combination of the following:

  1. a highly effective method of first choice = a method with a low failure rate (i.e. less than 1% per year) like sexual abstinence, combined oral contraceptives, implants, injectables, some Intra Uterine Devices (IUDs), vasectomized partner

     together with
  2. a method of second choice like condom, diaphragm, or cup pessary

Exclusion Criteria:

Criteria regarding gastrointestinal conditions:

* Short bowel syndrome
* Ileostomy, colostomy or rectal pouch
* Relapse during screening

Criteria regarding medical history:

* History of or existence of active tuberculosis
* History of or existence of urolithiasis
* History of or existence of human immune deficiency virus (HIV), Hepatitis B or C
* History of malignancy within the past five years (excluding basal cell carcinoma of the skin)
* Previous opportunistic infection
* History of serious drug sensitivity

Criteria regarding concomitant diseases:

* Significant cardiac arrhythmia, bradycardia or tachycardia or any other significant finding in the electrocardiogram (ECG)
* Congestive heart failure
* Uncontrolled arterial hypertension
* Uncontrolled asthma
* Renal disease
* Renal insufficiency defined as glomerular filtration rate (GRF) <50 ml/min/1.73 m² (estimated GRF according to Cockcroft-Gault)
* Psychiatric illness
* Known or suspected immunodeficiency
* Laboratory abnormalities: hemoglobin <8.5 g/dl, white blood cell count <3500/mm³, platelet count <125 000/mm³, clinically relevant elevation of liver enzymes, serum creatinine level >=1.4 mg/dl, hematuria (>=10 erythrocytes/field on dipsticks)

Criteria regarding concomitant circumstances:

* Pregnancy, lactation
* History of alcohol and/or drug dependence
* Heavy smoking (more than 20 cigarettes per day)
* Use of prohibited drugs or treatments
* Patient not able or not willing to follow study procedures due to physical or psychological limitations or language problems
* Participation in another investigational drug or vaccine trial within the last three months or concurrently with this study
* Vaccination with life attenuated viruses within 4 weeks prior to study start
* Patient with any medical condition which, in the opinion of the investigator or his designee, could jeopardize or compromise the ability of the patient to participate in the trial
* Patients possibly dependent on the investigator or the sponsor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of SC12267 (4SC-101) at a dose of 35 mg once daily in patients with Crohn's Disease (CD) or Ulcerative Colitis (UC) after a 12 week therapy as measured by the number of patients with complete or partial response. | after a 12 week therapy

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the safety and tolerability of SC12267 (4SC-101) at a dose of 35 mg once daily in patients with CD or UC and to explore plasma levels (trough values) of SC12267 (4SC-101). | after a 12 week therapy

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herrlinger, Prof., Principal Investigator — Robert Bosch Krankenhaus, Stuttgart, Germany
Locations (16):
- Bulgaria (3):
  - Tokuda Hospital Gastroenterology Division Internal Medicine Department, Sofia
  - UMHAT "Sv. Ivan Rilski" Gastroenterology Clinic, Sofia
  - UMHAT "Tsaritsa Ioanna" - ISUL Gastroenterology Clinic, Sofia
- Germany (10):
  - Charité, Universitätsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Klinikum der Ruhr-Universität Bochum, St. Josef-Hospital, I. Medizinische Klinik, Bochum
  - Universitätsklinikum Freiburg, Gastroenterologie, Hepatologie, Endokrinologie und Klinische Infektiologie, Freiburg im Breisgau
  - Schwerpunktpraxis für chronisch entzündliche Darmerkrankungen, Hamburg
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Technische Universität München II. Medizinische Klinik des Klinikums rechts der Isar, München
  - Gastroenterologische Gemeinschaftspraxis am Germania-Campus, Münster
  - Universitätsklinikum Regensburg Klinik und Poliklinik für Innere Medizin I, Regensburg
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
- Romania (3):
  - Elias University Emergency Hospital, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - University Emergency Hospital, Bucharest

REFERENCES:
- [Derived] Herrlinger KR, Diculescu M, Fellermann K, Hartmann H, Howaldt S, Nikolov R, Petrov A, Reindl W, Otte JM, Stoynov S, Strauch U, Sturm A, Voiosu R, Ammendola A, Dietrich B, Hentsch B, Stange EF. Efficacy, safety and tolerability of vidofludimus in patients with inflammatory bowel disease: the ENTRANCE study. J Crohns Colitis. 2013 Sep;7(8):636-43. doi: 10.1016/j.crohns.2012.09.016. Epub 2012 Oct 16. PMID 23078909
- [Derived] Kulkarni OP, Sayyed SG, Kantner C, Ryu M, Schnurr M, Sardy M, Leban J, Jankowsky R, Ammendola A, Doblhofer R, Anders HJ. 4SC-101, a novel small molecule dihydroorotate dehydrogenase inhibitor, suppresses systemic lupus erythematosus in MRL-(Fas)lpr mice. Am J Pathol. 2010 Jun;176(6):2840-7. doi: 10.2353/ajpath.2010.091227. Epub 2010 Apr 22. PMID 20413687